CLINICAL TRIAL: NCT01057472
Title: Repeatability and Feasibility of Infant Spirometry
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REK Vest 2009/1771
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Prematurity
Keywords: Repeatability of measurements
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Term born babies: Term born babies
- Preterm babies ready for discharge: Preterm babies ready for discharge
- Preterm stable babies 1500 grams: Preterm stable babies 1500 grams

SUMMARY:
This is a study examining repeatability and feasibility of a new method for measurement of lung function in babies. A flexible vest is placed around the torso of the baby, and changes in tidal volume and flow is measured. The study will enable a better understanding of the usefulness of this equipment in a neonatal intensive care unit. The equipment is made by VOLUSENSE Norway AS, and marketed under the name FloRight. The equipment is owned by Volusense Norway AS during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Being a Term born and preterm born babies

Exclusion Criteria:

* Being in an unstable clinical condition

Ages: 4 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term born and preterm born babies
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Repeatability of measurements performed by two different nurses before and after a meal in term babies (10), preterm babies before discharge (10) and preterm babies weighing approximately 1500 grams | Before and after a meal

SECONDARY OUTCOMES:
Feasibility of the measurements in the NICU | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Halvorsen, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Pediatric Department, NICU, Bergen, Norway

REFERENCES:
- See also: Related Info — http://www.volusense.com/Products.aspx